CLINICAL TRIAL: NCT05034003
Title: Clinical and Radiographic Performance of Zirconia and Composite Strip Crowns for Primary Incisors
Brief Title: Success of Zirconia and Composite Strip Crowns for Primary Incisors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zafer Cavit Cehreli, DDS, PhD, Prof.Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: anterior crown rest
Record Dates: First submitted 2021-08-24; First posted 2021-09-05 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Dental Caries in Children
Keywords: zirconia crowns, composite strip crowns, dental caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- zirconia crowns (Experimental): Zirconia crowns placed on primary incisor teeth
  Interventions: Device: Zirconia crown
- composite strip crowns (Experimental): composite strip crowns placed on primary incisor teeth
  Interventions: Device: composite strip crown
- Control tooth (No Intervention): Caries-free primary incisor tooth

INTERVENTIONS:
Device: Zirconia crown — Esthetic crowns for capping primary incisor with caries
  Arms: zirconia crowns
Device: composite strip crown — Esthetic resin restoration for primary incisor with caries
  Arms: composite strip crowns

SUMMARY:
The purpose of this study is to evaluate and compare the clinical and radiographic performance of zirconia and composite strip crowns bonded on primary incisors

DETAILED DESCRIPTION:
Zirconia and composite strip crowns will be placed on at least two primary incisor teeth, in a split mouth design. A caries-free primary incisor tooth will be used as control. 100 patients will be included in the study. The teeth will be randomized into two groups according to the crown type.

Group 1: Zirconia crown 2: Composite Strip Crown 3: Control tooth. Plaque index, gingival index, crown retention, presence of restoration failure, gingival margin extension, color match of the crowns and pulpal health of the teeth will be clinically evaluated at baseline and 1., 6., 12., 18., 24. months. The restorations will be evaluated radiographically at 6., 12. and 18. months. Intra-oral photos will be taken directly after treatment and at control appointments.

The data will be analysed statistically using Fisher's Exact Test and pearson's chi-square test; and Log-rank and the Kaplan-Meier will be used to estimate survival percentages.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parent of the patients who accept to participate and sign the informed consent
* Patients who have at least two primary maxillary incisor with caries that require crown restoration
* Teeth that have healthy lamina dura and periodontal ligament
* Teeth with no mobility and enough root length
* Patients that have good cooperation to the procedure

Exclusion Criteria:

* Patients and parent of the patients who don't accept to participate and sign the informed consent
* Teeth that are previously restored
* Patients who are uncooperative
* Teeth that doesn't have opposing primary incisors
* Patients who have bruxism or deep-bite
* Teeth that are close to be erupted
* Teeth that have vital or non-vital pulp therapy

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Number of zirconia and composite strip crowns that showed successful retention over two years | 2 years
  Long-term clinical success of zirconia and composite strip crowns placed on primary incisors

CONTACTS AND LOCATIONS:
Overall Officials: zafer c cehreli, Principal Investigator — Hacettepe university , Faculty of dentistry, ankara/Turkey
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)